CLINICAL TRIAL: NCT01839786
Title: Evaluation of Lung Doppler Signals in Pulmonary Hypertension
Status: Terminated | Type: Observational
Sponsor: Echosense Ltd. (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: DOP14
Record Dates: First submitted 2013-04-18; First posted 2013-04-25 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2013-04

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Doppler; Valsalva
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PHTN patients: 2. Patients who underwent RHC in the past and were diagnosed with PHTN (retrospective arm)

SUMMARY:
The purpose of this study is to evaluate the lung Doppler signals in patients with pulmonary hypertension that undergo (prospective arm) or underwent (retrospective arm) right heart catheterization (RHC) in order to assess whether this non-invasive tool could be used in pulmonary hypertension diagnosis and monitoring.

DETAILED DESCRIPTION:
PROTOCOL SUMMARY

Title: Evaluation of lung Doppler signals (LDS) in pulmonary hypertension (PHTN) Device: SONARA/tek transcranial Doppler (TCD) system Study Objectives: To evaluate the LDS in patients with PHTN that undergo (prospective arm) or underwent (retrospective arm) right heart catheterization (RHC) in order to assess whether these signals can be used in pulmonary hypertension diagnosis and monitoring.

Study Design:

Two study arms:

1. Prospective arm to measure LDS during right heart catheterization in patients undergoing the procedure for evaluation of PHTN.
2. Retrospective arm to measure LDS in patients in whom previous RHC confirmed the presence of PHTN.

Recruitment target: Prospective arm: 50 patients during 18 months. Retrospective arm: 50 patients during 18 months.

Study Population:

1. Patients suspected of PHTN by echocardiogram, who are scheduled to undergo RHC (prospective arm)
2. Patients who underwent RHC in the past and were diagnosed with PHTN (retrospective arm)

Study endpoint:

1. Comparison of pulmonary blood pressures at rest, following vasodilator medication and following upper extremities exercise as measured by RHC and by the LDS during the Valsalva maneuver.
2. Determining LDS characteristics of PHTN patients

ELIGIBILITY:
Inclusion Criteria:

1. Prospective arm:

   * Man or woman aged over 18.
   * With suspicion or diagnosis of pulmonary hypertension.
   * Scheduled to undergo right heart catheterization
   * Able and willing to give informed consent.
2. Retrospective arm:

   * Man or woman aged over 18.
   * With diagnosis of pulmonary hypertension confirmed by right heart catheterization in the past.
   * Able and willing to give informed consent.

Exclusion Criteria:

1. Both arms:

   * Minor (aged < 18).
   * People unable or unwilling to give informed consent.
   * Hemodynamically unstable patients.
   * Pregnant women.
2. Prospective arm only:

   * Patients with contra-indication to right heart catheterization.
   * Patients incapable of performing a Valsalva maneuver.
   * Patients with recent myocardial infarction, high degree AV block, severe aortic stenosis or glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of PHTN
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-05; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Find specific features that characterize lung signals of PHTN patients in comparison to control patients | 18 months
  The outcomes will be elaborate by statistical analysis of whole group data

CONTACTS AND LOCATIONS:
Overall Officials: Issahar Ben-Dov, MD, Principal Investigator — Sheba Medical center, Pulmonary institute
Locations (1):
- Sheba Medical Center, Pulmonology department, Ramat Gan, Israel